CLINICAL TRIAL: NCT01901692
Title: Randomized Trial Comparing Sorafenib and Transarterial Chemoembolization Plus External Beam Radiotherapy in Patients With Hepatocellular Carcinoma Showing Macroscopic Vascular Invasion
Brief Title: Sorafenib vs.TransArterial Chemoembolization Plus RadioTherapy in Hepatocellular Carcinoma With Macrovascular Invasion
Acronym: START
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Young-Suk Lim, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMC IRB 2013-0627
Record Dates: First submitted 2013-07-14; First posted 2013-07-17 (Estimated); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: Hepatocellular Carcinoma
Keywords: liver cancer; first-line; tumor thrombus; vascular invasion
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TACE+External beam RT (Experimental): Transarterial chemoembolization plus external beam radiation therapy
  Interventions: Radiation: TACE+External beam RT
- Sorafenib (Active Comparator): Sorafenib 800 mg/day orally
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Radiation: TACE+External beam RT — Trans-arterial chemoembolization (TACE) every 6 weeks + external beam radiation therapy starting within 3 weeks after first TACE
  Arms: TACE+External beam RT
Drug: Sorafenib — Sorafenib 800 mg/day orally
  Other Names: Nexavar
  Arms: Sorafenib

SUMMARY:
To evaluate and compare the efficacy and safety of sorafenib versus trans-arterial chemoembolization plus external beam radiation therapy in patients with hepatocellular carcinoma invading major intrahepatic vessels

DETAILED DESCRIPTION:
Current practice guidelines recommend only sorafenib for patients with hepatocellular carcinoma invading major intrahepatic vessels. However, recent data from observational studies suggest that the combination of transarterial chemoembolization and external beam radiotherapy would be as effective as sorafenib.

ELIGIBILITY:
Inclusion Criteria:

* Age >19 years
* Child-Pugh class A liver function
* Performance status: Eastern Cooperative Oncology Group (ECOG) score 0 or 1
* Hepatocellular carcinoma (HCC) confirmed by dynamic CT or MRI, or by biopsy
* HCC invasion of first or second branch portal vein or hepatic vein or inferior vena cava
* Reserved unilateral portal blood flow at least in partial
* HCC size larger than 1 cm and less than 50% of total liver volume
* No confirmed extrahepatic metastasis
* Adequate hematopoietic function Hemoglobin ≥ 8.5 g/dL Absolute neutrophil count ≥ 750/mm3 Platelet count ≥ 30,000/mm3
* Creatinine < 1.5mg/dL
* No plan for pregnancy or breast feeding. Active contraception.
* Willing to give informed consent

Exclusion Criteria:

* Prior history to or exposure of transarterial chemoembolization, external beam radiation to liver, or sorafenib
* Complete obstruction of hepatic outflow
* Confirmed extrahepatic metastasis of HCC
* HCC occupying more than 50% of liver volume
* Uncontrolled ascites of hepatic encephalopathy
* Prior liver transplantation
* Positive for human immunodeficiency virus (HIV)
* Active gastric or duodenal ulcer
* Other uncontrolled comorbidities or malignancy
* Inability to give informed consent

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2013-07-29 (Actual); Primary Completion 2017-01-20 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) rate | at 12 weeks after randomization
  Progression is defined as progressive disease (PD) by independent radiologic review according to RECIST criteria (version 1.1), termination of the assigned treatment, or death from any cause, assessed by Kaplan-Meier analysis and log-rank test for treatment comparisons with the intention-to-treat principle.

SECONDARY OUTCOMES:
Progression-free survival (PFS) rate | at 24 weeks and up to 4 years after randomization
  Progression is defined as progressive disease (PD) by independent radiologic review according to RECIST criteria (version 1.1), termination of the assigned treatment, or death from any cause, assessed by Kaplan-Meier analysis and log-rank test for treatment comparisons.
Radiologic response rate | at 12 and 24 weeks after randomization
  Radiologic response rate by independent radiologic review according to RECIST criteria (version 1.1), , assessed by Chi-square test or Fisher's exact test, as appropriate.
treatment-crossover rate | at 12 and 24 weeks after randomization
  Crossover of treatment is permitted after confirming the disease progression during the initially assigned treatment, assessed by Kaplan-Meier analysis and log-rank test for treatment comparisons.
time to progression | up to 4 years after randomization
  The median time to progression assessed by Kaplan-Meier analysis and log-rank test for treatment comparisons.
Overall patient survival rate | up to 4 years after randomization
  The median overall patient survival rate assessed by Kaplan-Meier analysis and log-rank test for treatment comparisons.
Exploratory analysis for overall patient survival rate | up to 4 years after randomization
  By using Cox proportional hazards model to evaluate the interaction between important baseline characteristics and the effect of treatments on overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Young-Suk Lim, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Yoon SM, Ryoo BY, Lee SJ, Kim JH, Shin JH, An JH, Lee HC, Lim YS. Efficacy and Safety of Transarterial Chemoembolization Plus External Beam Radiotherapy vs Sorafenib in Hepatocellular Carcinoma With Macroscopic Vascular Invasion: A Randomized Clinical Trial. JAMA Oncol. 2018 May 1;4(5):661-669. doi: 10.1001/jamaoncol.2017.5847. PMID 29543938